CLINICAL TRIAL: NCT06308094
Title: 320-detector Computed Tomography to Assess Myocardial Extracellular Volume Fraction in Patients With Atrial Fibrillation Before AF Ablation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00429859
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; ECV; Prognosis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Masking Description: Two independent blinded trained readers will detect, interpret and quantify interstitial fibrosis using CT images, to ascertain intra- and inter-observer variability. The readers will determine the region of interest (ROI), myocardial and blood pool attenuation values in the pre-contrast and 5 minutes delayed acquisition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afib with ECV measurement (Other): patients who are referred for catheter ablation will undergo additional CT acquisition for measurement of ECV to determine if there is any association between ECV expansion and Afib burden.
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — Pre-ablation CT is clinically acquired in patients undergoing catheter ablation. This study entails additional acquisition of the left ventricle to assess extracellular volume (ECV)

SUMMARY:
This study explores the relationship between myocardial fibrosis and patient outcomes in Atrial Fibrillation (AF), specifically after catheter ablation. It aims to use Cardiac CT, an accessible tool, to measure left ventricular extracellular volume (ECV) as an indicator of fibrosis. The study will assess if higher ECV levels correlate with increased risks of AF recurrence, hospitalization, and poor cardiac function recovery. Positive findings could make ECV a key factor in deciding AF treatment strategies.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the most common arrhythmia and is associated with significant healthcare-related expenses. With the aging population, the prevalence of AF is increasing. AF frequently co-exists with heart failure (HF) with reduced (HFrEF) or preserved (HFpEF) ejection fraction. The relationship between AF and HF is complex, and one condition constitutes a risk factor for the other. Myocardial interstitial fibrosis is a hallmark of myocardial remodeling occurring as a consequence of risk factor exposure leading to both AF and heart failure. However, the role of interstitial fibrosis in the prognosis of patients with atrial fibrillation with and without heart failure remains unknown.

AF has a significant impact on patients' well-being and quality of life. In addition to coping with uncomfortable symptoms, individuals with this condition face an increased risk of future adverse events like frailty, stroke, dementia, and all-cause mortality. To address these concerns, many patients opt for procedures such as AF ablation, hoping for a cure. While the results of this procedure show promise, a small percentage of patients who undergo AF ablation may experience a recurrence of the arrhythmia or find that the participant's heart's systolic function does not fully recover. The investigators aim is to investigate whether there is a connection between myocardial fibrosis and poor outcomes following AF ablation.

Cardiac MRI (CMR) has been the gold standard methodology of quantification of interstitial fibrosis. Diffuse interstitial fibrosis can be quantified by extracellular volume (ECV) imaging. CMR-based left ventricular ECV has been associated with adverse outcomes in multiple cardiovascular disease states. However, the availability of CMR is confined only to tertiary centers with expertise. Cardiac CT is an alternative way to detect and quantify interstitial fibrosis by quantification of ECV. CT-derived ECV has been shown in multiple studies to have an excellent correlation with CMR-derived ECV. Cardiac CT is widely available and has a higher spatial resolution. Since as part of the standard pre-ablation routine, patients will undergo a cardiac CT scan to accurately map the anatomy of the participant's heart, investigators ought to measure ECV parameters during this visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 21 years old at the time of enrollment.
* Patients must be able to give informed consent.
* Patients with symptomatic paroxysmal/persistent atrial fibrillation (AF).
* Eligible patients must be determined to be suitable candidates for ablation to treat AF by their cardiologist and/or electrophysiologists regardless of this protocol.
* Patients are scheduled to have a pre-procedure cardiac CT upon the discretion of their electrophysiologists

Exclusion Criteria:

* Known allergy to iodinated contrast media.
* Elevated serum creatinine (> 1.5mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula).
* Patients with a positive urine or serum pregnancy test will be excluded from this study.
* Patients with heart transplantation.
* Patients with polymorphic ventricular tachycardia (VT) or presenting in electrical storm.
* Presence of any other history or condition that the investigator feels would be problematic.
* Patient with iodinated contrast administration for other reason 24 hours prior to investigational CT.
* Patients who have a heart pacemaker, metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain, mechanical heart valves and prosthetics that contain metal.
* Patients with severe claustrophobia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation | Post procedure up to 90 days
  Patients will undergo computed tomography (CT) imaging with a total of 4 CT image acquisition (2 clinical and 2 research) During the follow-up visit with the primary electrophysiologist within 90 days after the procedure, the patient will be assessed for recurrence of atrial fibrillation.
Occurrence of ER visits, hospitalizations for cardiovascular causes | Post procedure up to 90 days
  Patients will be assessed for any emergency room visits, or hospitalizations for any cardiovascular causes.

SECONDARY OUTCOMES:
Change in Ejection Fraction | Post procedure up to 90 days
  As a follow-up measure, the patient will proceed to have an echocardiogram to check for improvement in ejection fraction. At the end of the study we we will analyze if there are any correlations between ECV expansion and lack of ejection fraction (EF) improvement.
Quality of Life as assessed by the Atrial Fibrillation Effect on Quality-of-Life (AFEQT) | Baseline, Post procedure up to 90 days
  Atrial Fibrillation Effect on Quality-of-Life will be used to measure quality of life. The score ranges from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Aronis, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code